CLINICAL TRIAL: NCT03162562
Title: Prospective Phase Ib Clinical Trial to Evaluate the Safety and Efficacy of Oregovomab and Hiltonol® as a Combinatorial Immunotherapy Strategy in Patients With Recurrent Advanced Epithelial Cancer of Ovarian, Tubal, or Peritoneal Origin
Brief Title: The Safety and Antitumor Activity of the Combination of Oregovomab and Hiltonol in Recurrent Advanced Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision to discontinue long-term follow-up
Sponsor: CanariaBio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QPT-ORE-003H
Record Dates: First submitted 2017-05-04; First posted 2017-05-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Cancer of Ovary; Neoplasms, Ovarian; Ovarian Cancer Stage IV; Ovarian Cancer Recurrent; Ovarian Cancer Stage III; Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — oregovomab; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oregovomab plus Poly ICLC (Hiltonol) (Experimental): Oregovomab Solution, 2 mg IV, every three weeks (weeks 0, 3, 6, and 9) and then once at week 16 plus poly ICLC Suspension, 2 mg IM, 30 minutes post-oregovomab infusion and 48 hours post-oregovomab infusion (total 10 doses)
  Interventions: Biological: Oregovomab; Drug: Poly ICLC

INTERVENTIONS:
Biological: Oregovomab — Monoclonal antibody against CA 125
Drug: Poly ICLC — Immune adjuvant
  Other Names: Hiltonol

SUMMARY:
This is a Phase Ib study to look at the combination of an antibody immunization vaccine strategy using oregovomab and an investigational stage immune booster (poly ICLC / Hiltonol), both of which have previously been used in combination with other cancer treatments and demonstrated to be active in advanced cancer, but which have not previously been used together. This study will assess the approach as to whether these two drugs can safely add to the response seen with either drug alone, both of which have doses that are based on prior studies.

Subjects with stable disease for whom a 12 week break from therapy for their persistent and progressive advanced ovarian cancer is appropriate, who have signed informed consent and for whom baseline clinical information is completed, will receive 4 cycles of oregovomab/Hiltonol immunization every three weeks (weeks 0, 3, 6, and 9). Blood will be obtained for to look for a CA125 specific T cell response at 12 weeks before initiating any additional therapy according to the best clinical judgment of the investigator. At week 16 the subjects will receive a final dose of the combination of oregovomab/Hiltonol and at week 17 will have an additional blood draw for analysis of T-cell response.

DETAILED DESCRIPTION:
This is a Phase Ib evaluation of the combination of an antibody immunization vaccine strategy using oregovomab and an investigational stage immune adjuvant (poly ICLC / Hiltonol), both of which have previously been used in combination with other cancer treatments and demonstrated to be bioactive in advanced cancer, but which have not previously been combined together. The doses selected for each agent have been selected previously through human clinical study for use in immunization protocols as a well-tolerated and bioactive immune stimulatory dose. For immunization purposes a maximum tolerated dose is not a relevant pharmacologic objective. Rather this is an exercise in efficiently assessing a preliminary immunization protocol as a cost effective product development strategy assessing the ability of the combination to safely augment the immune signals measurable with either agent alone, both of which have been titrated to the current dose based on the principle of bell shaped dose response in immunization in prior studies.

Subjects with stable disease for whom a 12 week break from cytotoxic therapy for their persistent and progressive advanced ovarian cancer is appropriate, who have signed informed consent and for whom baseline clinical information including laboratory, radiologic and physical documentation of their status is completed, will receive 4 cycles of oregovomab/Hiltonol immunization every three weeks (weeks 0, 3, 6, and 9). Blood will be obtained for the measurement of CA125 specific T cell immunity at 12 weeks before initiating continuing salvage therapy according to the best clinical judgment of the investigator. At week 16 the subjects will receive a final immunization with oregovomab/Hiltonol and at week 17 an additional blood draw for analysis of T-cell immunity.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects with CA125-associated, advanced ovarian cancer (FIGO Stage III/IV) previously treated and now presenting with recurrent or persistent disease.
2. Must have a histological diagnosis of epithelial adenocarcinoma of ovarian, tubal or peritoneal origin that is persistent or progressive following multiple rounds of prior standard of care and experimental therapy.
3. Must have had an elevated serum CA125 level twice the upper limit of normal (per reference lab normal range) measured within 4 weeks of enrollment.
4. Must have measurable disease by radiographic or physical criteria suitable for evaluation according to RECIST v1.1 for documentation of disease response or progression.
5. Must have a Functional Performance Status of less than or equal to 2 on the ECOG scale (Appendix VII).
6. Must have reached legal age to consent.
7. Must have medical assessment consistent with prognosis for an expected survival of at least 6 months and be clinically appropriate to receive a 12 week hiatus from any cytotoxic treatment according to the best clinical judgement of the treating investigator.
8. Must have voluntarily agreed to participate and have signed the informed consent, and are willing to complete all study procedures.

Exclusion Criteria:

1. Compromised hematopoietic function (hemoglobin <8.0 g/dL; lymphocyte count <300 mm3; neutrophil count <1000 mm3; platelet count <100,000 mm3).
2. Hepatic dysfunction defined as a bilirubin >1.5 times the upper normal limits, LDH, SGOT and SGPT>2 times upper limits of normal or albumin <3.5 g/dL.
3. Renal dysfunction defined as a serum creatinine >1.6 mg/dL.
4. Pregnant or breast-feeding. (While pregnancy is unlikely in view of the disease and previous surgery, subjects whom the investigator considers may be at risk of pregnancy will have a pregnancy [beta-HCG] test and will be using a medically approved contraceptive method).
5. Have an active autoimmune disease (e.g., rheumatoid arthritis, SLE, ulcerative colitis, Crohn's Disease, MS, ankylosing spondylitis) requiring continuing immune suppressive therapy.
6. Known allergy to murine proteins or have had a documented anaphylactic reaction to any drug, or a known hypersensitivity to diphenhydramine or other antihistamines of similar chemical structure.
7. Chronically treated with systemic doses of immunosuppressive drugs such as cyclosporin, ACTH, or corticosteroids.
8. Active infection causing fever.
9. Recognized immunodeficiency condition including cellular immunodeficiencies, hypogammaglobulinemia or dysgammaglobulinemia; subjects who have acquired, hereditary, or congenital immunodeficiencies, including HIV infection or have been splenectomized.
10. Uncontrolled diseases other than cancer will be excluded. Subjects with chronic diseases that are well controlled (e.g., diabetes mellitus, hypertension) are eligible.
11. Have received other investigational drugs within 30 days of enrollment.
12. Have contraindications to the use of pressor agents (e.g., SC epinephrine), notably monoamine oxidase inhibitor (MAOI) use.
13. Unable to read or understand, and/or unwilling to sign a written consent form which must be obtained prior to treatment.
14. Known to have recent history of drug abuse or alcoholism.
15. Have participated in a prior oregovomab clinical trial. Prior treatment with Hiltonol® does not exclude a subject from participation.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Change in laboratory values, physical findings (physical examination), vital signs, subjective patient experience and treatment-related adverse events as assessed by CTCAE v4.0 | Week 0 to Week17+30 days
  The primary outcome is to establish the preliminary safety regarding the combination of the anti-CA-125 monoclonal antibody oregovomab and the TLR3 agonist immune adjuvant poly ICLC (Hiltonol ®) as a strategy to induce CA125 specific anti-tumor immunity in heavily pretreated subjects with progressive ovarian cancer.

SECONDARY OUTCOMES:
Evaluation of cellular immune response to oregovomab. | Week 0, Week 12, Week 17
  Evaluation of the cellular immune response to oregovomab by a CA125 specific cellular immune response assay
Evaluation of human anti-mouse antibody (HAMA) response to oregovomab. | Week 0, Week 12, Week 17
  Evaluation of HAMA response to oregovomab by a commercial HAMA assay.
Time to overall survival | Up to Week 173
  Evaluation of overall survival up to three years after study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Nicodemus, MD FACP, Study Director — AIT Strategies
Locations (2):
- United States (2):
  - Florida Hospital Cancer Institute, Orlando, Florida
  - VCU Massey Cancer Center, Dalton Oncology Clinic, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicodemus CF, Wang L, Lucas J, Varghese B, Berek JS. Toll-like receptor-3 as a target to enhance bioactivity of cancer immunotherapy. Am J Obstet Gynecol. 2010 Jun;202(6):608.e1-8. doi: 10.1016/j.ajog.2009.12.001. Epub 2010 Jan 18. PMID 20080226